CLINICAL TRIAL: NCT05570916
Title: Zip-Stitch® in Minimally-Invasive Surgery (ZIMS) - Safety & Efficacy in Hysterectomy
Acronym: ZIMS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ZSX Medical LLC (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QD-PRO-054 Rev006; R44HD104539 (NIH)
Record Dates: First submitted 2022-10-04; First posted 2022-10-07 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Laparoscopic Hysterectomy
Keywords: Hysterectomy; Laparoscopic hysterectomy; minimally invasive hysterectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Test Article - Zip-stitch Clips (Experimental): Zip-stitch clips for vaginal cuff closure during laparoscopic hysterectomy
  Interventions: Device: Zip-stitch(R)
- Reference Group (Other): Will not be comparative against the test article, but will be performed for reference and safety.
  Interventions: Device: Reference suture

INTERVENTIONS:
Device: Zip-stitch(R) — Zip-stitch clips for vaginal cuff closure during laparoscopic hysterectomy
  Arms: Test Article - Zip-stitch Clips
Device: Reference suture — Standard suture for vaginal cuff closure during laparoscopic hysterectomy
  Other Names: V-Loc or VICRYL sutures
  Arms: Reference Group

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of the Zip-stitch® Vaginal Cuff Closure System. This will be primarily done by measuring the frequency of implant passing following system use. Also assessed will be relevant safety and efficacy endpoints as compared to a two-to-one reference group.

DETAILED DESCRIPTION:
This study is a prospective, blinded, randomized, controlled study to assess the safety and efficacy of the Zip stitch® System in maintaining vaginal cuff closure following minimally-invasive hysterectomy. Participating subjects will be randomized and evaluated for implant passing, successful cuff closure, healing, adverse events, dyspareunia, and pain. Blinded follow-up will involve in-person visits at one week and six weeks. There will be additional unblinded follow-up in person at six months post-operatively and by telephone at 12 months post operatively.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated Informed Consent Form 2. Stated willingness to comply with all study procedures, including participation in follow-up visits and telephonic follow-up 3. Female 18 years and older 5. Indicated for Laparoscopic Hysterectomy (includes Total Laparoscopic Hysterectomy, Laparoscopic Assisted Vaginal Hysterectomy, or robotic assisted vaginal hysterectomy)

Exclusion Criteria:

1. History of Human Immunodeficiency Virus (HIV)
2. History of Hepatitis C
3. History of diabetes that, in the opinion of the investigator, may delay healing
4. Current use of systemic corticosteroids
5. Active infection of genitals, vagina, cervix, uterus or urinary tract
6. Active bacteremia, sepsis or other active systemic infection
7. Presence of Sexually Transmitted Infection (STI)
8. Evidence of pelvic inflammatory disease (PID)
9. Known clotting defects or bleeding disorders
10. Hemoglobin < 8 g/dL
11. Metastatic disease
12. On anticoagulant therapy
13. Participation in another interventional trial
14. Pregnancy
15. Abnormal Papanicolaou test (PAP) results that have not been fully evaluated, or in the opinion of the investigator may indicate abnormal vaginal cuff healing
16. Co-morbidities that, in the opinion of the investigator, may indicate risk of abnormal vaginal cuff healing
17. Intra-operative: Bowel injury during laparoscopic hysterectomy procedure prior to attempted cuff closure
18. Intra-operative: Bladder injury during laparoscopic hysterectomy procedure prior to attempted cuff closure
19. Intra-operative: Cases in which surgeon cannot identify adequate tissue along the cuff to apply suture laparoscopically
20. Intra-operative: Cases requiring conversion to laparotomy prior to study intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
Safety: The primary safety endpoint in this study is frequency of vaginal cuff dehiscence. | This will be evaluated through six-weeks post-operative.
  Frequency of vaginal cuff dehiscence
Efficacy: The primary efficacy endpoint for this study is frequency of implant passing following cuff closure. | This will be evaluated through six weeks post operative.
  Frequency of implant passing

SECONDARY OUTCOMES:
Number of Participants With Successful Vaginal Cuff Closure | Performed at one week, six weeks, and six months after surgery
  Binary, visual surgeon cuff closure evaluation.
Number of Participants With Vaginal Cuff Healing | Performed at six weeks, and six months after surgery
  Binary, visual surgeon cuff healing evaluation.
Comparison of Number of Participants With Implant Passing - Test to Reference | Evaluated at six weeks and six months post-operative
  Percentage of subjects experiencing implant passing will be compared between test and reference groups.
Percentage of Participants With Implant Passing Events Determined to Impact Patient Safety | Evaluated through six-month follow-up
  Each reported implant passing event will be evaluated for association with adverse events. Compared as a percentage of patients in the test vs. reference groups.
Comparison of Incidence of Adverse Events - Test to Reference | Evaluated through six-month follow-up
  Adverse events and serious adverse events will be tabulated for both the test and reference groups.
Number of Participants With Non-increase in Dyspareunia at Follow-up | Evaluated through six-month follow-up
  Non-increase in reported individual subject dyspareunia from baseline to six month follow-up will be compared (test versus reference group) using the relevant sexual discomfort module of the Female Sexual Function Index (FSFI). The FSFI is a validated metric of female sexual function, where lower scores indicate poor sexual function. Non-increase in sexual discomfort will be compared between test and control groups.
Number of Participants With Non-increase in Pain at Follow-up | Evaluated through six-month follow-up
  Non-increase in reported individual subject pain from baseline to six-month follow-up will be compared (test versus reference group) using an 11-point Numerical Rating Scale, where 0 indicates no pain, and 10 indicates maximum possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: David Holtz, MD, Principal Investigator — Main Line Health
Locations (5):
- United States (5):
  - Northwestern University, Chicago, Illinois
  - Unified Women's Clinical Research, Winston-Salem, North Carolina
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - Tidewater Clinical Research, Virginia Beach, Virginia
  - Mon Health Medical Center, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ZSX Medical website — https://www.zsxmedical.com/